CLINICAL TRIAL: NCT00538200
Title: A Randomised Trial of Oral Nutritional Supplements Versus Dietary Advice on Clinical Outcomes in Patients With COPD
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) Nutrition Support Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ELIA002
Record Dates: First submitted 2007-09-04; First posted 2007-10-02 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Malnutrition
Keywords: Nutrition; COPD
MeSH Terms: conditions — Malnutrition; Pulmonary Disease, Chronic Obstructive | interventions — Dietary Supplements; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Dietary Advice
  Interventions: Other: Dietary Advice
- 2 (Other): Supplements
  Interventions: Dietary Supplement: Oral Nutritional Supplements (Fortisip)

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Supplements (Fortisip) — These products are classified as non-medicinal, borderline substances, foods for special medical purposes. A range of commercially available liquid oral nutritional supplements (Fortisip) will be offered daily for a 3 month period.
  Arms: 2
Other: Dietary Advice — Standard dietary advice
  Arms: 1

SUMMARY:
The purpose of this study is to determine the best form of dietary intervention to undernourished individuals with COPD.

The research aims to test the null hypothesis that there is no difference between oral nutritional supplements and dietary advice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age >18 years
* At risk of malnutrition
* Competent to provide written informed consent and able to answer questions
* Able to eat and drink
* Willingness to take part in the trial and to follow the trial protocol
* FEV1 <80% predicted and FEV1/FVC <0.7

Exclusion Criteria:

* Requirement for tube or parenteral nutrition
* Galactosemia
* Receiving current oral nutritional supplementation
* Palliative care
* Chronic renal disease requiring dialysis
* Liver failure
* Malignancy
* Participation in other studies
* Bronchiectasis
* Those already under the care of a dietitian

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2008-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is Quality of Life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marinos Elia, Professor, Principal Investigator — University of Southampton
Locations (1):
- Southampton University Hospitals NHS Trust, Southampton, Hampshire, United Kingdom